CLINICAL TRIAL: NCT01130701
Title: A Phase II Pilot Study to Evaluate the Efficacy and Safety of Neoadjuvant Chemoradiotherapy With Capecitabine, Panitumumab and External Beam Radiation, in Patients With Localized, Non-Metastatic Pancreatic Adenocarcinoma
Brief Title: A Pilot Study to Evaluate the Efficacy and Safety of Neoadjuvant Chemoradiotherapy With Capecitabine, . . .
Acronym: PMABIIS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never went beyond FDA application for an IND #. FDAA required institutional DSMC which this institution then lacked.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Bilal Piperdi, MD, University of Massachusetts Medical School
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UM2010-01
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2011-08

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Neoadjuvant; Panitumumab; Capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Panitumumab; Radiation; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Neoadjuvant capecitabine, panitumumab and radiation — Patients will receive six weekly doses of panitumumab (2.5mg/kg) in conjunction oral capecitabine 825 mg/m2 PO bid Mon-Friday and external beam radiation therapy. Panitumumab and oral capecitabine will begin on the first week of external beam radiotherapy and will continue throughout the course of external beam radiation therapy, and will be discontinued following the conclusion of external beam radiation therapy.
  Patients will be reevaluated for surgical resection 4-6 weeks after completion of neoadjuvant therapy.
  After surgical resection, adjuvant systemic chemotherapy with gemcitabine for six months is strongly recommended for all patients.
  Other Names: Xeloda; Vectibix; NSC # 742319

SUMMARY:
In this study, a new chemotherapeutic agent, panitumumab, will be tested in combination with another chemotherapeutic drug, capecitabine, along with external radiotherapy, to find out whether this combination is effective and safe to use before surgery.

DETAILED DESCRIPTION:
Surgical resection remains the standard procedure for patients with localized resectable pancreatic cancer.

Neoadjuvant or preoperative therapy with chemotherapy and radiation therapy has been proposed as an alternative approach in patients with localized pancreatic adenocarcinoma.

Advantages are: 1) early start of systemic therapy targeting micrometastatic disease; 2) increased compliance with chemoradiotherapy; 3) increase primary tumor complete resection rates; 4) avoidance of surgery in patients with rapidly developing metastatic disease; and 5) importantly, it provides an important resource for research in terms of tissue acquisition before and after therapy . Finally, this is an opportunity to test the safety and efficacy of a novel combination of weekly panitumumab, oral capecitabine and radiation in pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Cytological or histological confirmation of pancreatic adenocarcinoma is required.
2. Only patients with localized and apparently resectable, non-metastatic tumors are eligible. All patients must be staged with a chest X-ray or chest CT and abdominal and pelvic CT scan or MRI.

   One of the following radiological criteria must be met and recorded in chart by dedicated surgeon prior to enrollment.

   A)Localized, potentially resectable : 1) no evidence of tumor extension to the celiac axis, hepatic artery or superior mesenteric artery; 2) no evidence of tumor encasement or occlusion of superior mesenteric vein (SMV) or the SMV/portal vein(PV) confluence; 3) no evidence of visceral or peritoneal metastasis

   B)Borderline resectable: 1) no extra pancreatic disease, (2) the following possible tumor-vessel relationships: an SMV-PV confluence that can be reconstructed even if short segment venous occlusion is present; tumor abutment of the SMA of ≤180°; or short segment encasement of the hepatic artery amenable to resection and reconstruction.

   Patients with the following radiological criteria are NOT eligible:

   A) Locally advanced disease: (1) no extra pancreatic disease, (2) tumor encasement of the SMA or celiac axis defined as tumor involvement of >180° of the arterial circumference. B) Radiographic evidence of distant organ or peritoneal metastases.
3. Age > 18 years.
4. ECOG performance status 0 and 1.
5. Patient must have adequate hematological, renal and hepatic function defined as:

   WBC > 2,000 cells/mm3 ANC>1500 cells/mm3 Hemoglobin > 9.0 g/dL Platelets > 100,000 cells/mm3 Serum creatinine < 1.5 x upper limit of normal (UNL) or a calculated creatinine clearance of > 50 mL/min calculated by Cockcroft-Gault method Total bilirubin < 2.5 mg/dl AST < 3x upper limits of normal ALT < 3x upper limits of normal
6. Serum calcium and magnesium levels within limits of normal
7. Patients may not have any prior therapy for carcinoma of the pancreas, nor prior abdominal radiation therapy.

Exclusion Criteria:

1. Patients with any other malignancy within 5 years of study entry, except curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
2. Psychiatric illness which would prevent the patient from giving informed consent.
3. Serious medical illness which would limit anticipated survival to < 12 weeks.
4. Protocol treatment would pose significant risk to an unborn child. Pregnant women should not be enrolled, and women of child-bearing age should be strongly encouraged to practice effective birth control during and for six months after the trial. Non-pregnant and non-breast-feeding. Female participants of child-bearing potential must have a negative urine or serum pregnancy test prior to registration. Perimenopausal participants must be amenorrheic > 12 months to be considered not of childbearing potential. All patients (men and women) of reproductive potential must agree to use an effective method of birth-control while receiving study therapy and for six months after completion of therapy.
5. Inability to swallow medication. Patients should have adequate, unassisted oral intake.
6. Inability to hold still and cooperate during radiotherapy.
7. Prior history of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or any evidence of interstitial lung disease on baseline chest CT scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To estimate the 3 year progression-free survival of patients with localized, resectable pancreatic cancer | 2 Years
  To estimate the proportions of patients (with localized, resectable and borderline resectable, non-metastatic pancreatic adenocarcinoma) treated with the study regimen alive at 2-years from the date of registration.

SECONDARY OUTCOMES:
To estimate resection rate | 1 Year
  To determine the fraction of patients that proceed to planned surgery with the removal of primary tumor (R0/R1) following neoadjuvant therapy; estimate the overall survival in this patient population; evaluate the rate of R0, R1 and R2 resection (defined as per 6th edition of AJCC Cancer Staging Manual) in patients treated with neoadjuvant therapy; the overall response rate to chemoradiation therapy; the biomarker response to chemoradiation through evaluation of circulating CA19-9 levels; to evaluate the toxicity associated with this regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Piperdi, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Willett CG, Czito BG. Does adjuvant chemoradiation benefit patients who have undergone resection of pancreatic or periampullary cancer? Nat Clin Pract Gastroenterol Hepatol. 2008 Jul;5(7):364-5. doi: 10.1038/ncpgasthep1152. Epub 2008 May 27. No abstract available. PMID 18506163
- [Result] Meyer JJ, Willett CG, Czito BG. Is there a role for advanced radiation therapy technologies in the treatment of pancreatic adenocarcinoma? Future Oncol. 2008 Apr;4(2):241-55. doi: 10.2217/14796694.4.2.241. PMID 18407737
- [Result] Geer RJ, Brennan MF. Prognostic indicators for survival after resection of pancreatic adenocarcinoma. Am J Surg. 1993 Jan;165(1):68-72; discussion 72-3. doi: 10.1016/s0002-9610(05)80406-4. PMID 8380315
- [Result] Snady H, Bruckner H, Cooperman A, Paradiso J, Kiefer L. Survival advantage of combined chemoradiotherapy compared with resection as the initial treatment of patients with regional pancreatic carcinoma. An outcomes trial. Cancer. 2000 Jul 15;89(2):314-27. doi: 10.1002/1097-0142(20000715)89:23.0.co;2-v. PMID 10918161